CLINICAL TRIAL: NCT01501799
Title: A Multicenter, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Adapalene and Benzoyl Peroxide Topical Gel 0.1%/2.5% (Actavis Mid-Atlantic LLC) To Epiduo™ (Adapalene and Benzoyl Peroxide) Gel 0.1%/2.5% (Galderma Laboratories, L.P.) and Both Active Treatments to Topical Gel Placebo (Actavis Mid-Atlantic Llc) in the Treatment of Mild to Severe Acne Vulgaris
Brief Title: A Bioequivalence Study With Clinical Endpoints Comparing Adapalene and Benzoyl Peroxide Topical Gel 0.1%/2.5% (Actavis Mid-Atlantic LLC) To Epiduo™ (Adapalene and Benzoyl Peroxide) Gel 0.1%/2.5% (Galderma Laboratories, L.P.) in the Treatment of Mild to Severe Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Actavis Mid-Atlantic LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACTA/ADAP/BP/2010
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Acne Vulgaris
Keywords: acne; adapalene/benzoyl peroxide; Epiduo; Mild to severe acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Benzoyl Peroxide; Gels; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adapalene 0.1% and benzoyl peroxide 2.5% topical gel (Experimental)
  Interventions: Drug: adapalene 0.1% and benzoyl peroxide 2.5% topical gel
- EPIDUO™ (adapalene 0.1% and benzoyl peroxide 2.5%) Gel (Active Comparator)
  Interventions: Drug: EPIDUO
- Vehicle Gel (Placebo Comparator)
  Interventions: Drug: Placebo (Vehicle Gel)

INTERVENTIONS:
Drug: adapalene 0.1% and benzoyl peroxide 2.5% topical gel — Dosage form: topical gel Dosage: A pea-sized amount was applied to each affected area of the face Frequency: once daily in the evening Duration: 12 weeks
  Arms: Adapalene 0.1% and benzoyl peroxide 2.5% topical gel
Drug: EPIDUO — EPIDUO (adapalene 0.1% and benzoyl peroxide 2.5%) Gel
  Arms: EPIDUO™ (adapalene 0.1% and benzoyl peroxide 2.5%) Gel
Drug: Placebo (Vehicle Gel) — Vehicle Gel
  Arms: Vehicle Gel

SUMMARY:
EPIDUO™ (adapalene and benzoyl peroxide) Gel 0.1%/2.5%, marketed by GALDERMA LABORATORIES, L.P., is a safe and effective topical therapy used for the treatment of acne vulgaris. Actavis Mid-Atlantic LLC has developed a generic formulation of adapalene and benzoyl peroxide topical gel 0.1%/2.5%,and the current study is designed to evaluate the safety and efficacy of this formulation to determine if it is bioequivalent to EPIDUO™.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant female patients must be between the ages of 12 and 40 years old inclusive.
2. Patients who are 18 years of age or older must have provided IEC/IRB approved written informed consent. Patients between the ages of 12 to 17 years of age must have provided IEC/IRB approved written assent; this written assent must be accompanied by an IEC/IRB approved written informed consent from the patient's legally acceptable representative (i.e., parent or guardian). In addition, all patients or their legally acceptable representatives (i.e., parent or guardian) must sign a HIPAA authorization, if applicable.
3. Patients must have a definite clinical diagnosis of mild to severe acne vulgaris (Grade 2, Grade 3 or Grade 4 on the IGE).
4. Patients must have a minimum of 20 inflammatory lesions and a maximum of 100 and a minimum of 25 and a maximum of 100 non-inflammatory lesions (i.e., open and closed comedones) and no more than 2 nodulocystic lesions (i.e., nodules and cysts) at baseline. For the purposes of study treatment and evaluation, these lesions should be limited to the facial treatment area. Lesions involving the eyes, angles of the nose (i.e., the lines around your nostrils and under the nostrils) and scalp should be excluded from the count. Patients may have acne lesions on other areas of the body (e.g., on the back).
5. Female patients of childbearing potential must have been using accepted methods of birth control or must agree to continue to practice abstinence, from 30 days prior to study entry to 30 days after the last administration of study drug. All female patients are considered to be of childbearing potential unless they have been surgically sterilized or have been postmenopausal for at least 1 year. Abstinence is an acceptable method of birth control. Any of the following methods of birth control are acceptable: oral contraceptives, contraceptive patches/implants (e.g., Norplant®) Depo-Provera®, double barrier methods (e.g., condom and spermicide) or IUD. Female patients must have a negative urine pregnancy test at baseline. A negative result of a pregnancy test having a minimum sensitivity of at least 50 mIU/ml for hCG should be obtained.
6. All male patients must agree to use accepted methods of birth control with their partners, from the day of the first dose administration to 30 days after the last administration of study drug. Abstinence is an acceptable method of birth control. Any of the following methods of birth control are acceptable: oral contraceptives, contraceptive patches/implants (e.g., Norplant®), Depo-Provera®, double barrier methods (e.g., condom and spermicide) or IUD.
7. Patients must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits.
8. Patients must be willing to refrain from using any other treatments for acne vulgaris, including antibiotics, other than the investigational product, for acne present on the face. Patients may use other topical acne treatments that do not have significant or measurable systemic absorption for treatment of acne of the back, shoulders and chest (e.g., benzoyl peroxide, salicylic acid).
9. Patients must be in good health and free from any clinically significant disease.
10. Patients who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to not change make-up brand/type or frequency of use throughout the study.

Exclusion Criteria:

1. Female patients who are pregnant, nursing or planning to become pregnant during study participation (Visit 1 through Visit 5) will be excluded from study participation.
2. Patients who have a known hypersensitivity to benzoyl peroxide, adapalene, and other retinoids, or their excipients will be excluded from study participation.
3. Patients who have conditions that may interfere with the evaluation of acne vulgaris. Such conditions include, but are not limited to the following lesions on the face: rosacea; seborrheic dermatitis; perioral dermatitis; corticosteroid-induced acne or folliculitis; carcinoid syndrome; squamous cell carcinoma; mastocytosis; acneiform eruptions caused by make-up or medication; bacterial folliculitis; facial psoriasis; and facial eczema.
4. Patients who have acne congoblata, acne fulminans, and secondary acne (e.g., chloracne and drug induced acne) will be excluded from participation.
5. Patients who have been treated with systemic antibiotics or systemic anti-acne drugs or systemic anti-inflammatory drugs within 30 days prior to baseline will be excluded from study participation.
6. Patients who have been treated with prescription and/or over-the-counter topical medications for the treatment of acne vulgaris including antibiotics, topical corticosteroids, α-hydroxy/glycolic acid, benzoyl peroxide, or topical anti-inflammatory medications on the face within 14 days prior to baseline will be excluded from study participation.
7. Patients who are currently taking or have been treated with systemic corticosteroids (including intranasal and inhaled corticosteroids) within 30 days prior to baseline will be excluded from study participation.
8. Patients who have started hormonal therapy or changed the dosage of their hormonal therapy within 3 months prior to baseline will be excluded from study participation. The dosage and frequency of use of any hormonal therapy started greater than 3 months prior to baseline must remain unchanged throughout the study (Visit 1 through Visit 5). Hormonal treatments include, but are not limited to, estrogenic and progestational agents such as birth control pills.
9. Patients who use androgen receptor blockers (such as spironolactone or flutamide) will be excluded from study participation.
10. Patients who have received oral retinoids (e.g., isotretinoin) within 180 days prior to study entry,or have used therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed) within 180 days prior to study entry, or have applied topical retinoids (e.g., tretinoin, tazarotene, adapalene) to the face within the 2 weeks prior to baseline will be excluded from study participation.
11. Patients who have received radiation therapy and/or anti-neoplastic agents within 90 days prior to baseline will be excluded from study participation.
12. Patients who have unstable medical disorders that are clinically significant or life-threatening diseases will be excluded from study participation.
13. Patients who have on-going malignancies requiring systemic treatment will be excluded from study participation. In addition, patients who have any malignancy of the skin of the facial area will be excluded from study participation.
14. Patients who have facial hair will be excluded from study participation. Unacceptable facial hair includes, but is not limited to, beards, and long side-burns. A well-trimmed mustache is acceptable. Patients who have performed wax epilation of the face within 14 days prior to baseline will also be excluded from study participation.
15. Patients who engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold, will be excluded from study participation.
16. Patients who consume excessive amounts of alcohol (greater than two drinks per day) or use drugs of abuse (including, but not limited to, cannabinoids and cocaine) as judged by history will be excluded from study participation.
17. Patients who have participated in an investigational drug study (i.e., patients have been treated with an investigational drug) within 30 days prior to baseline will be excluded from study participation. Patients who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion.
18. Patients who have been previously enrolled in this study will be excluded from study participation.
19. Patients who have had within 30 days prior to baseline or during the study cryodestruction or chemodestruction, dermabrasion, photodynamic therapy, acne surgery, intralesional steroids, or x-ray therapy will be excluded from study participation.
20. Patients who have had laser therapy, and electrodessication to the facial area within 180 days prior to study entry will be excluded from participation.
21. Patients who have had cosmetic procedures (e.g., facials) which may affect the efficacy and safety profile of the investigational product within 14 days prior to study entry will be excluded from participation.
22. Patients who have had general anesthesia for any reason and patients who have received neuromuscular blocking agents within 14 days prior to study entry will be excluded from study participation.
23. Patients who have a baseline local irritation score of 3 (severe, marked/intense) as scored using the Application Site Reaction Scale (Section 5.2) will be excluded from participation.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 885 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percent change in inflammatory and non-inflammatory lesions from Baseline to Week 12 | Week 12
  The mean percent change from Baseline to Visit 5 (End of Treatment) in the inflammatory and non-inflammatory lesion counts.
Treatment-emergent adverse events | 12 Weeks
  All adverse events (AEs) and treatment-emergent AEs reported during the study were summarized for the safety assessment. A treatment-emergent AE was defined as any event not present prior to the initiation of treatment with the investigational products or any event present at Baseline that worsened in either intensity or frequency following exposure to investigational products.
Signs and Symptoms of Local Irritation | 12 Weeks
  Patients will be evaluated for any signs and/or symptoms as separate scores of local irritation, including: erythema, dryness, burning / stinging, erosion, edema, pain, scaling, and itching using the following scale:
  0 = None
  1. = Mild, barely perceptible
  2. = Moderate, distinctive presence
  3. = Severe, marked/intense

SECONDARY OUTCOMES:
The proportion of "success" patients at Visit 5 using the IGE | 12 Weeks
  The proportion of "success" patients at Visit 5 using the IGE, where "success" was defined as a two-grade improvement.
Mean Percent Change in Total Lesion Count from Baseline to Visit 5 | 12 Weeks
  The mean percent change in the total lesion count from Baseline to Visit 5.

CONTACTS AND LOCATIONS:
Overall Officials: Nagashayana G., M.D., Study Director — Lotus Labs Pvt Ltd; Nermina Nakas, M.D., M.P.H., Study Director — Jubilant Clinsys, Inc
Locations (25):
- United States (8):
  - Center for Dermatology Clinical Research Inc., Fremont, California
  - FXM Research Corp., Miami, Florida
  - FXM Research Miramar, Miramar, Florida
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Adult & Pediatric Dermatology, Overland Park, Kansas
  - Skin Search of Rochester Inc., Rochester, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Haber Dermatology and Cosmetic Surgery Inc., South Euclid, Ohio
- FXM Research International - Belize, Belize City, Belize District, Belize
- India (16):
  - Raga's Skin Care, Bangalore, Bangalore
  - MS Clinical Research Pvt. Ltd., Bangalore, Bangalore
  - Chamarajpet Skin and Laser Centre, Chamarajpet, Bangalore
  - Rajbal Polyclinic & Research Center, Kalyan Nagar, Bangalore
  - Department of Skin & STD, Kempegowda Institute of Medical Sciences,, V.V. Puram, Bangalore
  - Bhagwan Mahaveer Jain Hospital, Vasanthnagar, Bangalore
  - Skin & Cosmetology Clinic, Banjara Hills, Hyderabad
  - Department of Dermatology, Durga Bai Deshmukh Hospital, Vidyānagar, Hyderabad
  - Bhatia Skin, Laser & Cosmetic Center, Anand Bazar, Indore
  - Swarnakar Super Specialty Centre, Anand Bazar, Indore
  - Skin Clinic, RNT Marg, Indore
  - Agrawal Skin & Laser Centre, Vijayanagar, Indore
  - Sri Gayathri Skin Care & Hair Transplant Centre, Dwarakanagar, Visakhapatnam
  - Dayal Clinic, Visakhapatnam, Visakhapatnam
  - B.V. Department of Dermatology King George Hospital, Visakhapatnam, Visakhapatnam
  - Skin & Cosmetology, Visakhapatnam, Visakhapatnam